CLINICAL TRIAL: NCT06095284
Title: Prescribing Trends and Associated Outcomes of Antiepileptic Drugs and Other Psychoactive Medications in US Nursing Homes Surrounding the COVID-19 Pandemic
Brief Title: Prescribing Trends and Associated Outcomes of Antiepileptic Drugs in US Nursing Homes Surrounding the COVID-19 Pandemic
Status: Enrolling by invitation | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: HM20025382; R01AG074358 (NIH)
Record Dates: First submitted 2023-10-19; First posted 2023-10-23 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Dementia
Keywords: Mood-stabilizing AED's; Nursing Home
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All nursing home residents included in the 2009-2021 MDS: All nursing home residents included in the 2009-2021 MDS
  Interventions: Other: Pre-Extraction Phase; Other: Extraction Phase; Other: Post-Extraction Phase
- Nursing home and non-nursing home residents diagnosed with an AD/ADRD condition: Nursing home and non-nursing home residents diagnosed with an AD/ADRD condition
  Interventions: Other: Pre-Extraction Phase; Other: Extraction Phase; Other: Post-Extraction Phase

INTERVENTIONS:
Other: Pre-Extraction Phase — This intervention requires the following procedures: Submitting data use agreement, MDS request defined and developed, Part D request, CMS public use file request defines and develop questionnaire
Other: Extraction Phase — Procedures include: Access VRDC for 2 years, Crosswalk CMS files and MDS using ID's, Preliminary analysis for validity/accuracy, Request revision/resubmission, Linked dataset created in VRDC and Distribute Questionnaire
Other: Post-Extraction Phase — Procedures include: De-identified data securely stored, analysis, dissemination and knowledge translation

SUMMARY:
Since the "National Partnership to Improve Dementia Care" debuted in 2012, almost all long-stay psychoactive prescribing has been graded by CMS, which has correlated to decreased use. However, some national data suggest that while these psychoactive medications are being used less, prescriptions of mood-stabilizing antiepileptic drugs (AEDs) have increased. Unlike all other psychoactive medications, AEDs prescribed in nursing homes are not mandatorily reported to CMS or graded in a quality-measure.

DETAILED DESCRIPTION:
Pilot studies from Virginia suggest increases in AEDs are concentrated entirely in dementia patients with no diagnosis of epilepsy and as a purposeful unmonitored alternative to antipsychotics. AEDs are not FDA approved for dementia symptoms, have weak efficacy evidence, and convey serious risk. Increasingly it seems likely that the Partnership's debut was an inflection point where the trend towards unmonitored alternative drugs for dementia symptoms sharply increased. Early Commonwealth data hints that the COVID pandemic represents a second critical point of inflection where the existing transition towards non-superior but unreported drugs is again rapidly accelerating. All outcomes associated with this evolving prescribing phenomenon remain unknown. That said, pilot data suggests that harms may be increasing without benefit, a development with relevance to all invested in improving dementia care including patients, caregivers, and policy makers.

ELIGIBILITY:
Inclusion Criteria:

* All long-stay nursing home residents will be included. We define long-stay nursing home residents as all individuals residing in a nursing facility place of service for more than 100 days
* All nursing home clinicians prescribing psychoactive drugs will be included.

Exclusion Criteria:

* Limited to nursing home residents with continuous fee-for-service or Medicare Advantage plans as well as continuous Part D coverage.
* Residents without continuous fee-for-service insurance (less than 3 percent of nursing home population) will be excluded.
* Less than 0.2% of nursing home residents are children; still, this study will be restricted to those > 21 years of age.
* Nursing home residents who are discharged before the end of the quarterly study periods will also be excluded.
* Residents with discharges for acute hospitalizations followed by facility reentry on the same record will not be excluded.
* Non-prescribing clinicians and clinicians that do not prescribe psychoactive medications will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will only include de-identified data sets that are eligible for download and analysis and that meet the inclusion and exclusion criteria. Only those 21 years or older will be included.
Sampling Method: Non-Probability Sample
Enrollment: 22500000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Quarterly rate of use and mean dose of AEDs in US nursing homes | The years 2009 to 2021
  Quarterly rate of use and mean dose of AEDs in US nursing homes 2009-2021

SECONDARY OUTCOMES:
Quarterly rate of use of AEDs in US nursing homes for long-stay residents | The years 2009 to 2012
  Quarterly rate of use of AEDs in US nursing homes for long-stay residents with and without: dementia, seizure-epilepsy, psychiatric diagnoses, neuropathic pain, an appropriate diagnosis for AED use
Quarterly rate of adverse health events among US nursing home residents prescribed or not prescribed AEDs | The years 2009 to 2021
  Quarterly rate of adverse health events among US nursing home residents prescribed or not prescribed AEDs from 2009 to 2021.
  Adverse health events include:
  * Detrimental nursing home outcomes including falls, cognitive scores, functional scores, harmful behaviors, weight loss, hospice, death
  * ER encounters (per 1000 nursing home days)
  * Hospitalizations (per 1000 nursing home days), potentially avoidable hospitalizations, medication related hospitalizations, costs of hospital care.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Winter, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States